CLINICAL TRIAL: NCT02991729
Title: Use of a Novel Decision Aid for Prenatal Aneuploidy Screening
Brief Title: Use of a Novel Computerized Decision Aid for Prenatal Aneuploidy Screening
Acronym: DAAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-1745
Record Dates: First submitted 2016-12-08; First posted 2016-12-13 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2018-01

CONDITIONS: Aneuploidy; Pregnancy Complications
Keywords: Decision aid
MeSH Terms: conditions — Aneuploidy; Pregnancy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine care (Active Comparator): These patients will receive routine care at our institution for counseling on aneuploidy screening; they will be counseled by a genetic counselor on options, and following counseling, will select their test of choice. All patients will complete a knowledge and demographics questionnaire prior to genetic counseling. Patients in this arm will then complete a knowledge and decisional conflict survey immediately following genetic counseling.
  Interventions: Other: Genetic counseling appointment
- Experimental (Experimental): These patients will use an iPad-based decision aid explaining options for aneuploidy screening and testing. They will then immediately be counseled by a genetic counselor on their options as is routine at our institution, and following counseling, will select their test of choice. All patients will complete a knowledge and demographics questionnaire prior to genetic counseling. Patients in this arm will then complete a knowledge and decisional conflict survey following use of the decision aid, and again immediately following genetic counseling.
  Interventions: Other: iPad-based decision aid; Other: Genetic counseling appointment

INTERVENTIONS:
Other: iPad-based decision aid — This is a novel decision aid developed by genetic counselors and Maternal Fetal Medicine physicians. It is used via an iPad and is interactive. It is available in English and Spanish has been piloted by 20 English and Spanish speaking women. It takes approximately 15 minutes to complete.
  Arms: Experimental
Other: Genetic counseling appointment — All participants will undergo an approximately 15 minute educational genetic counseling appointment regarding aneuploidy screening options. Should family history concerns be identified on intake, this visit may be extended to include a discussion of additional issues.

SUMMARY:
The investigators aim to assess whether use of a novel, tablet-based computerized decision aid for aneuploidy screening is similar to routine care with a brief genetic counseling visit in improving patient knowledge and decreasing decisional conflict.

DETAILED DESCRIPTION:
184 women will be randomized in a 1:1 fashion to use of a novel computerized iPad-based decision aid in addition to routine counseling or routine counseling only during a single study visit. This decision aid was developed at a 10th grade literacy level using input from Maternal Fetal Medicine physicians and certified genetic counselors, and piloted by 20 English and Spanish speaking women of varying education levels. Following completion of genetic counseling, participants will complete several surveys assessing knowledge and decision conflict. Data will be abstracted regarding demographics, screening and diagnostic testing uptake, and testing results.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy at less than 22 weeks gestation
* English or Spanish speaking
* Undergoing genetic counseling at North Carolina Women's Hospital for aneuploidy screening

Exclusion Criteria:

* Known fetal anomalies
* Known multiple gestations
* Prior genetic counseling or aneuploidy screening in current pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2018-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Carlson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.

REFERENCES:
- [Derived] Carlson LM, Harris S, Hardisty EE, Hocutt G, Vargo D, Campbell E, Davis E, Gilmore K, Vora NL. Use of a novel computerized decision aid for aneuploidy screening: a randomized controlled trial. Genet Med. 2019 Apr;21(4):923-929. doi: 10.1038/s41436-018-0283-2. Epub 2018 Sep 14. PMID 30214066

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: These patients will use an iPad-based decision aid explaining options for aneuploidy screening and testing. They will then immediately be counseled by a genetic counselor on their options as is routine at our institution, and following counseling, will select their test of choice. All patients will complete a knowledge and demographics questionnaire prior to genetic counseling. Patients in this arm will then complete a knowledge and decisional conflict survey following use of the decision aid, and again immediately following genetic counseling.
  iPad-based decision aid: This novel decision aid was developed by genetic counselors and Maternal Fetal Medicine physicians. It is used via an iPad and is interactive. It is available in English and Spanish has been piloted by 20 English and Spanish speaking women. It takes approximately 15 minutes to complete.
  Genetic counseling appointment: All participants will undergo an approximately 15-min educational genetic counseling appointment
Period: Overall Study
Arm/Group | Routine Care | Experimental
Started | 105 | 92
Completed | 105 | 92
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Knowledge score (on 12 point scale) for each participant will be analyzed by group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Care | Experimental | Total
Number analyzed (Participants) | 105 | 92 | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (5.7) | 32.7 (5.6) | 32.6 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 92 | 197
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 63 | 47 | 110
  Black | 19 | 10 | 29
  Hispanic/Latino | 15 | 24 | 39
  Asian | 5 | 9 | 14
  Unspecified/other | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Knowledge Score
Description: All patients in the intervention arm will complete a knowledge questionnaire following completion of the decision and and again immediately following genetic counseling. The investigators will assess noninferiority of the decision aid on participant knowledge, with primary outcome comparing knowledge after completion of the decision aid in the intervention arm, to knowledge following genetic counseling only in the routine care arm. The questionnaire is a modification of the validated Maternal Serum Screening Knowledge Questionnaire. This is on a 12-point scale (values 0-12), with higher score indicating greater knowledge.
Time Frame: At completion of genetic counseling for the Routine Care Group and at completion of decision aid and genetic counseling for Experimental Group, approximately 10-60 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Routine Care | Experimental
Number analyzed (Participants) | 105 | 92
score on a scale | 10.6 (1.9) | 10.2 (2.4)
Statistical Analysis 1: Comparison: Routine Care vs Experimental; Test type: Non-Inferiority — The non-inferiority limit was 1 point on the questionnaire scale; p = 0.929, Wilcoxon rank-sum — a priori threshold for statistical significance was p<0.05

2. Secondary Outcome: Decisional Conflict Score
Description: A low-literacy decisional conflict questionnaire will be used. This will be completed by patients in the intervention arm following use of the decision and and again following genetic counseling. It will be completed by patients in the routine care arm following genetic counseling. Decisional conflict at all time points will be compared - specifically, decisional conflict following decision aid completion in the Experimental Group will be compared to decisional conflict following genetic counseling in the Routine Care Group, and decisional conflict following both decision aid completion and genetic counseling in the Experimental Group will be compared to decisional conflict following genetic counseling in the Routine Care Group. This questionnaire is on a 40 point scale (values 0-40), with higher score indicating higher level of decisional conflict.
Time Frame: At completion of decision aid (Experimental group) and completion of genetic counseling (all participants), approximately 10-60 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Routine Care | Experimental
Number analyzed (Participants) | 105 | 92
score on a scale
  Pre-genetic counseling/post-decision aid | NA (NA) — This group did not complete a decisional conflict score prior to genetic counseling. | 1.6 (3.5)
  Post-Genetic Counseling | 1.7 (4.8) | 0.2 (3.5)
Statistical Analysis 1: Comparison: Routine Care vs Experimental; Decisional conflict was measured in 2 separate time points in the experimental group - both prior to and following genetic counseling. This analysis compares decisional conflict in the routine care group (after counseling only) to the experimental group following decision aid completion but prior to genetic counseling (first row, second column in above table); Test type: Superiority; p = 0.369, Wilcoxon rank-sum
Statistical Analysis 2: Comparison: Routine Care vs Experimental; Decisional conflict was measured in 2 separate time points in the experimental group - both prior to and following genetic counseling. This analysis compares decisional conflict in the routine care group (after counseling only) to the experimental group following decision aid completion and genetic counseling (second row, second column in above table); Test type: Superiority; p = 0.003, Wilcoxon rank-sum
Statistical Analysis 3: Comparison: Experimental; Decisional conflict was measured in 2 separate time points in the experimental group - both prior to and following genetic counseling. This analysis compares decisional conflict pre-genetic counseling/post-decision aid to post-genetic counseling; Test type: Superiority; p = 0.003, Wilcoxon signed-rank

3. Secondary Outcome: Test Chosen
Description: For participants in the intervention arm, initial choice of aneuploidy screening following use of the decision aid will be compared to final test chosen following genetic counseling.
Time Frame: At completion of decision aid and at completion genetic counseling, approximately 10-60 minutes
Population: Some participants chose not to answer this question and so the numbers above reflect the number of participants for whom we have data.
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: Pre-genetic Counseling; Experimental: Post-genetic Counseling: These patients will use an iPad-based decision aid explaining options for aneuploidy screening and testing. They will then immediately be counseled by a genetic counselor on their options as is routine at our institution, and following counseling, will select their test of choice. All patients will complete a knowledge and demographics questionnaire prior to genetic counseling. Patients in this arm will then complete a knowledge and decisional conflict survey following use of the decision aid, and again immediately following genetic counseling.
  iPad-based decision aid: This novel decision aid was developed by genetic counselors and Maternal Fetal Medicine physicians. It is used via an iPad and is interactive. It is available in English and Spanish has been piloted by 20 English and Spanish speaking women. It takes approximately 15 minutes to complete.
  Genetic counseling appointment: All participants will undergo an approximately 15-min educational genetic counseling appointment
Arm/Group | Experimental: Pre-genetic Counseling | Experimental: Post-genetic Counseling
Number analyzed (Participants) | 85 | 67
Participants
  None/US only | 17 | 11
  First trimester screen | 35 | 28
  Cell free DNA | 27 | 25
  Quadruple analyte screen | 3 | 2
  Chorionic villus sampling | 0 | 1
  Amniocentesis | 1 | 0
  Don't know | 2 | 0

4. Secondary Outcome: Supplementary Tests Performed
Description: Use of additional aneuploidy screening or testing modalities (cell-free DNA, chorionic villus sampling, or amniocentesis in addition to initial screening test) in the current pregnancy will be assessed up to 22 weeks gestation.
Time Frame: 22 weeks gestation
Population: This analysis was updated to include only invasive testing - these numbers represent those women undergoing chorionic villus sampling or amniocentesis for high risk screening results.
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Care | Experimental
Number analyzed (Participants) | 4 | 2
Participants
  Invasive testing for high-risk results | 2 | 1
  No invasive testing for high-risk results | 2 | 1

ADVERSE EVENTS:
Time Frame: Over the course of the study visit, approximately 1 hour
Description: Patients were encouraged to contact study PI and given contact information for any questions or concerns.
Arm/Group | Routine Care | Experimental
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/92
Other Adverse Events (participants affected / at risk) | 0/105 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT02991729/Prot_SAP_000.pdf